CLINICAL TRIAL: NCT01309802
Title: A 28-Day Randomized, Double-Blind, Placebo-Controlled Clinical Trial and 5-Year Prospective Outcomes Study: A Two-Part Study of BOTOX® Therapy for Ischemic Digits
Brief Title: A Two-Part Study of BOTOX® Therapy for Ischemic Digits
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-SIUSOM-11-001
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Raynaud's Disease
Keywords: botox; raynaud's; botulinum toxin; botulinum toxin A; raynaud's disease; raynaud's syndrome; raynaud's phenomenon; ischemic digits; ischemia; botox treatment; onabotulinum; onabotulinum toxin; onabotulinum toxin type A
MeSH Terms: conditions — Raynaud Disease; Ischemia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (No Intervention): no intervention
- onabotulinum toxin type-A (Active Comparator): up to 4 injections per hand dosage per injection: 100 units diluted in 2.0 mL normal saline; dosing will not exceed 360 units in a 3 month interval frequency: no less than 28 days between injections duration: during Study Year 1
  Interventions: Drug: onabotulinum toxin type-A

INTERVENTIONS:
Drug: onabotulinum toxin type-A — up to 4 injections per hand dosage per injection: 100 units diluted in 2.0 mL normal saline; dosing will not exceed 360 units in a 3 month interval frequency: no less than 28 days between injections duration: during Study Year 1
  Other Names: BOTOX®; botulinum toxin type A
  Arms: onabotulinum toxin type-A

SUMMARY:
Treating patients with Raynaud's phenomenon who have chronic pain and ulcerations is extremely challenging. Published reports and our previous work support our hypothesis that symptomatic patients experience relief of pain and healing of ulcerations with minimal adverse effects when treated with botulinum toxin type A (Btx-A) injections for Raynaud's phenomenon. The proposed study is the first clinical trial and prospective study designed to document whether or not 1) Btx-A injection relieves pain in a patient's hand affected with Raynaud's disease better than a placebo within 28 days of injection, and 2) Btx-A injection relieves pain associated with Raynaud's disease for longer than 28 days, improving patients' quality of life. Through this study we intend to further determine the effect of injected Btx-A on relieving chronic pain and ulcerations to the ischemic hand while characterizing the patients for whom this treatment is most effective.

DETAILED DESCRIPTION:
PROJECT SUMMARY OVERVIEW: Treating patients with Raynaud's phenomenon who have chronic pain and ulcerations is extremely challenging. Pharmacologic vasodilators and surgical sympathectomies offer variable benefits. Case reports, small retrospective outcomes studies, and our previous work documenting symptomatic patients treated with botulinum toxin type A (Btx-A) injections for Raynaud's phenomenon have demonstrated relief of pain and healing of ulcerations with minimal adverse effects. We propose to conduct the first clinical trial and prospective study documenting the efficacy of this novel treatment modality.

STUDY AIMS: The aims of this proposal are to 1) examine the short-term efficacy of Btx-A injection compared to placebo in treating pain associated with digit ischemia due to Raynaud's disease, and 2) describe the long-term efficacy of Btx-A injection in treating pain associated with digit ischemia due to Raynaud's disease by measuring patient satisfaction and quality of life changes over time.

APPROACH: Two groups of patients will be enrolled: Group 1 will consist of patients with primary Raynaud's disease (n=20) and Group 2 of patients with secondary Raynaud's (n=20). Comparisons between treatment (Btx) and placebo (saline) will occur during the first 28 days to determine Btx-A's short-term efficacy. Follow-up visits will occur at Days 7 and 28. Post-assessment on Day 28 marks the beginning of the longitudinal observational study of patient outcomes. Placebo will no longer be used and patients still suffering from pain will be eligible for additional Btx-A injections. Patients may receive up to 4 injections of Btx-A during the 1-year study period if pain or ulcerations recur. During the study period participants will be followed to collect data on pain-free intervals, ulcer healing, subsequent treatment choices, patient satisfaction, and changes in quality of life and hand function. Group comparisons will be made to analyze results. Further stratifications for data analysis will be made as enrollment numbers allow to control for additional demographic and disease variables. Quality-adjusted life-years will be calculated to help determine the societal and individual cost of this treatment.

HYPOTHESIS: We hypothesize that 1) Btx-A injection relieves ischemic pain associated with Raynaud's disease better than a placebo within 28 days of injection, and 2) Btx-A injection relieves ischemic pain associated with Raynaud's disease for longer than 28 days, improving patients' quality of life. Through this study we intend to further elucidate the efficacy of injected Btx-A on relieving chronic pain and ulcerations to the ischemic hand while characterizing the patients for whom this treatment is most effective. This data will help us to apply for national funding to become the coordinating center for a multi-center clinical trial. The results of this research have enormous potential to impact millions of patients who suffer with Raynaud's phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-75 years
* diagnosed with Raynaud's disease/phenomenon
* ischemia not due to peripheral artery disease or other vascular disease
* otherwise healthy individual
* up-to-date tetanus immunization
* ability to return/be available for follow-up evaluations
* ability/willingness to give informed consent

Exclusion Criteria:

* HIV/AIDS positive or otherwise immunocompromised
* history of neuromuscular disease
* reported allergy to BOTOX®; reported allergy to lidocaine or other local anesthetic agent
* ever received botulinum toxin vaccine
* ultrasound or angiogram showing digital ischemia due to blocked vessel and not Raynaud's disease
* history or symptoms of any significant medical problem in the last year (i.e., bradycardia, impaired cardiovascular function, liver disease)
* symptoms of infection or illness during initial enrollment
* pregnant or lactating women
* unable or unwilling to maintain abstinence or use contraception for 28 days following all injections
* cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05; Primary Completion 2016-05-19 (Actual); Study Completion 2016-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Neumeister, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing data.

REFERENCES:
- [Background] Neumeister MW. Botulinum toxin type A in the treatment of Raynaud's phenomenon. J Hand Surg Am. 2010 Dec;35(12):2085-92. doi: 10.1016/j.jhsa.2010.09.019. PMID 21134617
- [Background] Neumeister MW, Chambers CB, Herron MS, Webb K, Wietfeldt J, Gillespie JN, Bueno RA Jr, Cooney CM. Botox therapy for ischemic digits. Plast Reconstr Surg. 2009 Jul;124(1):191-201. doi: 10.1097/PRS.0b013e3181a80576. PMID 19568080
- [Background] Sycha T, Graninger M, Auff E, Schnider P. Botulinum toxin in the treatment of Raynaud's phenomenon: a pilot study. Eur J Clin Invest. 2004 Apr;34(4):312-3. doi: 10.1111/j.1365-2362.2004.01324.x. No abstract available. PMID 15086364
- [Background] Van Beek AL, Lim PK, Gear AJL, Pritzker MR. Management of vasospastic disorders with botulinum toxin A. Plast Reconstr Surg. 2007 Jan;119(1):217-226. doi: 10.1097/01.prs.0000244860.00674.57. PMID 17255677
- [Background] Fregene A, Ditmars D, Siddiqui A. Botulinum toxin type A: a treatment option for digital ischemia in patients with Raynaud's phenomenon. J Hand Surg Am. 2009 Mar;34(3):446-52. doi: 10.1016/j.jhsa.2008.11.026. PMID 19258141
- See also: U.S. Food and Drug Administration — http://www.fda.gov/Drugs/default.htm
- See also: Drugs@FDA; U.S. Food and Drug Administration — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Onabotulinum Toxin Type-A
Started | 25 | 23
Completed | 13 | 14
Not Completed | 12 | 9

BASELINE CHARACTERISTICS:
Population: Race and Ethnicity were not collected for this protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Onabotulinum Toxin Type-A | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 19 | 42
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Full Range); unit: years] | 53.3 [24 to 73] | 49.2 [26 to 70] | 51.3 [24 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patient Reported Pain-free Days
Description: Subjective pain scales [visual analogue scale (VAS) and faces pain assessment]. Subjects reporting total number of pain free days within the time period of 0-28 days.
Time Frame: baseline to 28 days
Measure: Number; unit: percentage of pain free days
Arm/Group | Placebo | Onabotulinum Toxin Type-A
Number analyzed (Participants) | 25 | 23
percentage of pain free days | 12 | 48

2. Secondary Outcome: Pain Related Quality of Life
Description: SF-12v2® Health Survey - Pain Enhanced
Time Frame: change from baseline to 28 days
Population: Data were not collected,
Arm/Group | Placebo | Onabotulinum Toxin Type-A
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Hand Function
Description: Quick-DASH (Disabilities of the Arm, Shoulder, and Hand) Outcome Measure
Time Frame: baseline to 28 days
Population: Data were not collected
Arm/Group | Placebo | Onabotulinum Toxin Type-A
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Patient Satisfaction
Description: The Optum SF-12v2® Health Survey - A Short Patient Reported Survey Measuring Health Using Excellent, Very Good, Good, Fair and Poor Indicators. On a scale from Excellent to Poor, Excellent being the maximum outcome. Good is scored as average. Patient satisfaction assessed as the percentage of participants who responded; Excellent, Very Good and Good on the health survey on average feeling between baseline and 28 days.
Time Frame: baseline to 28 days
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Onabotulinum Toxin Type-A
Number analyzed (Participants) | 25 | 23
percentage of participants | 12 | 48

5. Secondary Outcome: Tissue Perfusion
Description: Doppler perfusion imager and Periscan image analysis software
Time Frame: baseline to 28 days
Population: Data were not collected
Arm/Group | Placebo | Onabotulinum Toxin Type-A
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: EQ-5D A Standardised Patient Reported Measure of Health Status for Clinical and Economic Appraisal
Description: A combined reported score measuring 5 dimensions; mobility, self care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels; no problems, some problems, extreme problems
Time Frame: baseline to 28 days
Population: not were not collected
Arm/Group | Placebo | Onabotulinum Toxin Type-A
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: For adverse events were followed to resolution.
Arm/Group | Placebo | Onabotulinum Toxin Type-A
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 5/25 | 2/23
Other Adverse Events (participants affected / at risk) | 25/25 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Onabotulinum Toxin Type-A (N=23)
Broken bone (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Collapsed Lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Throat Swelling (General disorders) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Onabotulinum Toxin Type-A (N=23)
Pain, Redness, Bleeding (General disorders) | 14 (35) | 14 (31)
Swelling, Tenderness, Bruising (General disorders) | 12 (17) | 7 (9)
Temporary Weakness or numbness of muscle (Musculoskeletal and connective tissue disorders) | 16 (32) | 11 (20)
Dizziness, Drowsiness (General disorders) | 3 (3) | 3 (4)
Dry Eyes, Dry Mouth (General disorders) | 1 (2) | 0
Vision Changes (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Increased Cough, Runny nose (General disorders) | 1 (2) | 0 (0)
Allergic Reaction or Itching (General disorders) | 2 (2) | 0 (0)
Tingling (General disorders) | 0 (0) | 1 (1)
Shortness of breath (General disorders) | 1 (1) | 2 (2)
Difficulty Swallowing (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes